CLINICAL TRIAL: NCT03928938
Title: Follow-up of Cancer Patients Receiving Immune Checkpoint Inhibitor Therapy by Electronic Patient Reported Outcomes-tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Koivunen, principal investigator, associate professor, Oulu University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9/2017
Record Dates: First submitted 2019-01-29; First posted 2019-04-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic follow-up (Experimental): Follow-up of cancer patients treated with immune checkpoint inhibitor therapy using electronic patient reported outcomes-tool
  Interventions: Device: Electronic patient reported outcomes

INTERVENTIONS:
Device: Electronic patient reported outcomes — Electronic patient reported outcomes-tool

SUMMARY:
Electronic patient reported outcome (ePRO) tools have improved survival and quality of life (QoL) of cancer patients receiving chemotherapy, and in the follow-up of lung cancer patients. Current study investigates electronic patient reported outcome tool in the follow-up of cancer patients receiving immune checkpoint inhibitor therapy.

Current study aims to evaluate 1) patient reported symptoms and their severity, 2) Number of triggered alerts by the tool and their correlation to treatment side-effects, cancer progression, other medical events or survival, 3) Correlation between different symptoms and the correlation of symptoms to treatment side-effects, cancer progression, other medical events or survival,4) QoL of patients and correlation of changes in QoL to treatment side-effects, cancer progression, other medical events or survival, 5) Patient compliance, 6) Correlation of baseline laboratory values to treatment side-effects, cancer progression, other medical events or survival.

DETAILED DESCRIPTION:
Please see the Brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Advanced cancers
3. Immune checkpoint inhibitor therapy initiated within +/- 2wks
4. Age >18y
5. ECOG 0-3
6. Patient compliant with the study procedures

Exclusion Criteria:

1. Immune checkpoint inhibitor therapy initiated > 2wks ago
2. General vulnerability affecting the participation in the trial
3. No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the spectrum of patient reported symptoms | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Percentages of patient reported symptoms using KaikuHealth 17 symptom e-questionnaire. Individual questions evaluate the presence of a specific symptom e.g. nausea. Questions are answered yes or no.
Change in Patient reported symptom severity | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Percentages of patient reported symptoms and their severity according NCI-CTCAE by KaikuHealth algorithm
Change in the number of triggered alerts by the tool | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Number of triggered alerts by the tool and their correlation to treatment side-effects, cancer progression, other medical events in percentages or survival.
Changes in Quality of Life according to QLQ-C30 Summary scores | At baseline, and at 4, 8, and 12weeks
  The correlation of the Summary score of QLQ-C30 to treatment side-effects, cancer progression, or other medical events or survival.
  The Core Quality of life questionnaire (QLQ-C30) is a validated cancer health-related quality-of-life questionnaire that includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality of life and financial impact. Subjects respond on a four-point-scale from "not at all" to "very much" for most items. Raw scores are linearly converted to a 0-100 scale. For the functioning scales and global QoL higher scores indicate better functioning; for the symptom scales higher scores indicate higher symptom burden. The summary score of QLQ-C30 is calculated from the mean of 13 of 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included).
Correlation between changes in different symptoms and their severity to treatment side-effects, cancer progression, other medical events, or survival. | At 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation between different patient reported symptoms and their severity to treatment side-effects, cancer progression or other medical events in percentages or survival.
Changes in Patient compliance Questionnaire | At 4, 8, and 12weeks
  Patient compliance using KaikuHealth e-questionnaire addressing usability (easiness to use from scale: very easy to very difficult; need of assistance to use the program: yes/no; how understandable are questions in symptom questionnaire from scale: totally agree to totally disagree) and user experience (use of the ePRO tool will better your cancer care: yes-no, do not know; use of the ePRO tool has been useful: yes-no-do not know; would you recommend the ePRO tool for cancer care: yes-no-do not know). Analysis is done on percentages of each answer choice at specific time point(s).
Changes in patient compliance according to answering rate to symptom questionnaires | At 4, 8, and 12weeks
  Patient compliance using response rates (within one week) to symptom questionnaires in percentages from sent requests
Change in patient compliance according to answering rates to QLQ-C30 questionnaire | At 4, 8, and 12weeks
  Patient compliance using response rates to QLQ-C30 questionnaires (within one week) in percentages from sent requests. The QLQ-C30 questionnaire includes five function domains (physical, emotional, social, role, cognitive), eight symptoms (fatigue, pain, nausea/vomiting, constipation, diarrhea, insomnia, dyspnea, and appetite loss), as well as global health/quality of life and financial impact. Subjects respond on a four-point-scale from "not at all" to "very much" for most items. Raw scores are linearly converted to a 0-100 scale. For the functioning scales and global QoL higher scores indicate better functioning; for the symptom scales higher scores indicate higher symptom burden. The summary score of QLQ-C30 is calculated from the mean of 13 of 15 QLQ-C30 scales (the Global Quality of Life scale and the Financial Impact scale are not included).
Correlation of change in baseline Hb values compared to control Hb values to treatment side-effects, cancer progression, other medical events or survival. | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation of change in baseline Hb values compared to control Hb values at specific timepoints to treatment side-effects, cancer progression, other medical events or survival.
Correlation of change in baseline leucocyte values compared to control leucocyte values to treatment side-effects, cancer progression, other medical events or survival. | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation of change in baseline leucocyte compared to control leucocyte values at specific timepoints to treatment side-effects, cancer progression, other medical events or survival.
Correlation of change in baseline lymphocyte values compared to control lymphocyte values to treatment side-effects, cancer progression, other medical events or survival. | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation of change in baseline lymphocyte values compared to control lymphocyte values at specific timepoints to treatment side-effects, cancer progression, other medical events or survival.
Correlation of change in baseline neutrophil values compared to control neutrophil values to treatment side-effects, cancer progression, other medical events or survival. | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation of change in baseline neutrophil values compared to control neutrophil values at specific timepoints to treatment side-effects, cancer progression, other medical events or survival.
Correlation of change in baseline CRP values compared to control CRP values to treatment side-effects, cancer progression, other medical events or survival. | At Baseline, and at 2-3, 4-5, 6-7, 8-9, and 11-12weeks
  Correlation of change in baseline CRP values compared to control CRP values at specific timepoints to treatment side-effects, cancer progression, other medical events or survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jussi P Koivunen, M.D., Ph.D, Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - Docarates Cancer Center, Helsinki
  - Pia Vihinen, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iivanainen S, Ekstrom J, Virtanen H, Kataja VV, Koivunen JP. Electronic patient-reported outcomes and machine learning in predicting immune-related adverse events of immune checkpoint inhibitor therapies. BMC Med Inform Decis Mak. 2021 Jun 30;21(1):205. doi: 10.1186/s12911-021-01564-0. PMID 34193140
- [Derived] Iivanainen S, Alanko T, Vihinen P, Konkola T, Ekstrom J, Virtanen H, Koivunen J. Follow-Up of Cancer Patients Receiving Anti-PD-(L)1 Therapy Using an Electronic Patient-Reported Outcomes Tool (KISS): Prospective Feasibility Cohort Study. JMIR Form Res. 2020 Oct 28;4(10):e17898. doi: 10.2196/17898. PMID 33112242

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03928938/Prot_SAP_000.pdf